CLINICAL TRIAL: NCT03071484
Title: Evaluation of the Efficacy of Transcranial Direct Current Stimulation in the Treatment of Cognitive Symptomatology in the Early Stages of Psychosis: Study Protocol of a Double-blind Randomized Controlled Trial
Brief Title: Efficacy of Transcranial Direct Current Stimulation in Treatment of Cognitive Deficits in Early Stages of Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Bairral de Psiquiatria (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Acioly Luiz Tavares de Lacerda, PhD, Instituto Bairral de Psiquiatria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2155/08
Record Dates: First submitted 2017-02-13; First posted 2017-03-07 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia
Keywords: Early Stages of Psychosis; Schizophrenia; Transcranial Direct Current Stimulation; Cognitive Symptomatology; Double-blind Randomized Controlled Trial
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Direct Current Stimulation (Experimental): After being randomly allocated, the experimental group will receive a 20 minutes of active 2-mA tDCS once a day on 10 consecutive weekdays.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham - tDCS (Placebo Comparator): The control group will receive a sham stimulation, which chosen parameters consists in after 40 seconds of real stimulation (2 mA), only a small current pulse occurred every 550 msec (110 mA over 15 msec) through the remainder of the 20-minute period.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — The tDCS is a non-invasive neuromodulatory technique that delivers low-intensity, direct current to cortical areas facilitating or inhibiting spontaneous neuronal activity.

SUMMARY:
Background: Cognitive deficits are a core symptom of schizophrenia even at the early stages of psychosis. To date, there has been reliable evidence that cognitive deficits are associated with outcomes in schizophrenia and early treatment could help to reduce the prominent disabling cognitive symptomatology which most schizophrenia patients still experience persistently. Outcomes in studies of repetitive transcranial magnetic stimulation in schizophrenia patients suggest the possibility that application of transcranial direct-current stimulation (tDCS) with inhibitory stimulation over the left temporo-parietal cortex and excitatory stimulation over the left dorsolateral prefrontal cortex could affect positive and negative symptoms, respectively. Positive effects of tDCS have also been reported on cognitive symptoms. The present study protocol hypothesis is that the development and utilization of potentially effective neuroenhancement tools such as a non-invasive brain stimulation technique like tDCS for the treatment and rehabilitation of cognitive impairment in early stages of Schizophrenia may contribute to the elucidation of the nature of the complex and dynamic processes in the brain during the early stages of the disease, and may lead to a better outcome.

Objectives: The aim of the present study protocol is to evaluate the efficacy of tDCS in the treatment of cognitive symptomatology in the early stages of psychosis.

Methods: Sixty patients in the early stages of psychosis will be randomly allocated to receive 20 minutes of active 2-mA tDCS or sham stimulation once a day on 10 consecutive weekdays. The anode will be placed over the left dorsolateral prefrontal cortex and the cathode over the left temporo-parietal cortex. Neuropsychological and psychiatric assessments will be performed at the time of consent (baseline), at 1 and 3 months following the end of the intervention (maintenance effect).

DETAILED DESCRIPTION:
The design of the present study protocol is a double-blind placebo controlled randomised clinical trial.

After being randomly allocated, the experimental group will receive a 20 minutes of active 2-mA tDCS once a day on 10 consecutive weekdays. The control group will receive a sham stimulation (placebo), which chosen parameters consists in after 40 seconds of real stimulation (2 mA), only a small current pulse occurred every 550 msec (110 mA over 15 msec) through the remainder of the 20-minute period.

Neuropsychological and psychiatric assessments will be performed at the time of consent (baseline), and at 1 and 3 months following the end of the intervention (maintenance effect). The primary outcome will be cognitive function and the second outcomes will be the positive and negative symptoms. Outcome assessments will be performed by trial research staff. Primary and second outcomes assessors (neuropsychologists and psychiatrists) and patients will be blinded to randomized allocation after assignment to interventions.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria include:

1. subjects of both gender, diagnosed with schizophrenia in early stage psychosis (first five years of illness), confirmed through the Structured Interview of the American Psychiatric Association Diagnostic and Statistical Manual of Mental Disorders - 4th edition (SCID-IV);
2. aged 17-60 years;
3. minimum of 4 years of schooling;
4. Intelligent Quotient (IQ) from low average to higher scores (IQ>70);
5. and the subjects should be receiving stable doses of antipsychotics for at least four weeks (antipsychotic dose stability criterion).

Exclusion Criteria:

1. presence of a history of cranioencephalic trauma with loss of consciousness with a time greater than 5 minutes;
2. history of central nervous system diseases that affect the brain;
3. unstable clinical conditions;
4. current diagnosis of substance abuse;
5. history of substance dependence in the last 6 months, except nicotine addiction;
6. current diagnosis of another Axis I condition, confirmed through SCID-IV.

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
MCCB™ MATRICS™ (Measurement and Treatment Research to Improve Cognition in Schizophrenia) Consensus Cognitive Battery | 3 months follow up
  A consensus cognitive battery for measuring cognition in schizophrenia,

SECONDARY OUTCOMES:
Positive and Negative Symptoms Scale (PANSS) | 3 months follow up
  Positive and Negative Symptoms Scale (PANSS)

CONTACTS AND LOCATIONS:
Overall Officials: Rabanea-Souza, MsC, Principal Investigator — Federal University of São Paulo
Locations (1):
- Laboratory of Interdisciplinary Clinical Neurosciences, Department of Psychiatry, Federal University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rabanea-Souza T, Cirigola SMC, Noto C, Gomes JS, Azevedo CC, Gadelha A, Cordeiro Q, Dias AM, Lacerda ALT. Evaluation of the efficacy of transcranial direct current stimulation in the treatment of cognitive symptomatology in the early stages of psychosis: study protocol for a double-blind randomized controlled trial. Trials. 2019 Apr 5;20(1):199. doi: 10.1186/s13063-019-3288-5. PMID 30953544